CLINICAL TRIAL: NCT02245711
Title: Intrathecal Autologous Mononuclear Cell Therapy for Limb Girdle Muscular Dystrophy
Brief Title: Cell Therapy in Limb Girdle Muscular Dystrophy
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Neurogen Brain and Spine Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NGBSI-12
Record Dates: First submitted 2014-09-12; First posted 2014-09-22 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Limb Girdle Muscular Dystrophy
Keywords: Limb Girdle Muscular Dystrophy; Autologous Bone Marrow Mononuclear cell therapy; Stem Cell
MeSH Terms: conditions — Muscular Dystrophies, Limb-Girdle

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stem Cell (Experimental)
  Interventions: Biological: Stem Cell

INTERVENTIONS:
Biological: Stem Cell

SUMMARY:
The purpose of this study was to study the effect of stem cell therapy on Limb Girdle Muscular Dystrophy patients.

ELIGIBILITY:
Inclusion Criteria:

* age group of 15 years-60 years
* limb girdle muscular dystrophy diagnosed on the basis of clinical presentation
* Electromyographic and Nerve Conduction velocity findings

Exclusion Criteria:

* presence of respiratory distress
* presence of acute infections such as Human Immunodeficient Virus/Hepatitis B Virus/Hepatitis C Virus
* malignancies
* acute medical conditions such as respiratory infection, fever, hemoglobin less than 8, bleeding tendency, bone marrow disorder, left ventricular ejection fraction < 30%
* pregnancy or breastfeeding

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2010-12; Primary Completion 2015-01 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in Functional Independence Measure (FIM) scale | 1 year
  Functional Independence Measure scale assesses the patients ability to carry out activities of daily living. At the follow up of 1 year, every patient in this study will be reevaluated on this scale.

SECONDARY OUTCOMES:
Change in Manual Muscle Testing (MMT) | 1 year
  Manual muscle testing is a procedure for the evaluation of the function and strength of individual muscles and muscle groups based on the effective performance of a movement in relation to the forces of gravity and manual resistance. On the follow up after 1 year, every patient will be reassessed on MMT to record changes in their muscle strength after stem cell therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Neurogen brain and spine institute, Navi Mumbai, Maharashtra, India